CLINICAL TRIAL: NCT02030444
Title: Randomized Study Comparing Standard Staging of Lung Cancer With Extended Staging Including EBUS-TBNA and PET-MRI
Brief Title: Extensive Staging in Lung Cancer
Acronym: ExtStaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to difficulties with recruiting
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ExtStaging-2014.1
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Lung Neoplasms
Keywords: Neoplasms Staging; Bronchoscopy; Nuclear Medicine; Radiology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard diagnostic work-up (No Intervention): All patients will undergo todays' standard work-up (examination for diagnosing and staging) of lung cancer. This will be individualized for each patient according to current guidelines.
- Extensive diagnostic work-up (Experimental): All patients will in addition to standard diagnostic work-up undergo PET-MRI and systematic mediastinal and hilar lymph node mapping using EBUS-TBNA (endobronchial ultrasound transbronchial needle aspiration of lymph nodes).
  Interventions: Procedure: PET-MRI and EBUS-TBNA

INTERVENTIONS:
Procedure: PET-MRI and EBUS-TBNA
  Arms: Extensive diagnostic work-up

SUMMARY:
The overall aim of this study is to compare standard staging of lung cancer (which includes clinical examination, CT, MRI, bone scan and PET-CT) with comprehensive staging - which includes the new staging methods (PET-MRI and systematic mapping of mediastinal and hilar lymph nodes using endobronchial ultrasound) with respect to disease stage and outcomes of therapy.

DETAILED DESCRIPTION:
The trial is a randomized, explorative study. Patients undergoing examinations for suspicions of lung cancer (Stage I-III) are randomized to either standard diagnostic work-up for lung cancer (Arm A, n=75) or comprehensive diagnostic work-up (Arm B, n=75) with standard examinations plus endobronchial-screening for metastatic lymph nodes (EBUS-TBNA) and PET-MRI.

All patients will undergo todays' standard examination for diagnosing and staging lung cancer. This will be individualized for each patient according to current guidelines. In addition to the standard diagnostic work-up, patients in the interventional group (ArmB) will undergo

1) PET-MRI 2) systematic mediastinal and hilar lymph node mapping using EBUS-TBNA (endobronchial ultrasound transbronchial needle aspiration of lymph nodes)

1. PET-MRI PET-MRI will be done immediate after the standard PET-CT using the same infusion of tracer (18-fluorodeoxyglucose, FDG). The sequence protocols used for MRI will be standardized for the study, according to each body compartment. Measurement of Standard Uptake Values (SUV) of the tracer (FDG) will be recorded in pathological lesions. In the mediastinum, each lymph node station will be evaluated with description of visible nodes.
2. Systematic mediastinal mapping The EBUS-TBNA will be done at the initial bronchoscopy and using standard conscious sedation according to the local guidelines at St.Olavs Hospital. Each lymph node station (station 2, 4, 7, 10 and 11 bilateral) will be examined and all lymph nodes ≥ 0,5 cm in short diameter that is easily accessible will be punctured for rapid on-site cytological evaluation (ROSE).

After the initial diagnostic work-up is completed, the patient will be given treatment according to existing guidelines for lung cancer based on the given clinical stage.

For patients undergoing surgery all accessible lymph nodes will be resected according to standard practice. Every resected lymph node will be carefully named according to the standard lymph station for comparison with clinical findings.

ELIGIBILITY:
1. Patients undergoing examinations on suspicion of lung cancer (both SCLC and NSCLC) at St. Olavs Hospital
2. Potentially curable disease at the referral time (Stage I-III, based on the first CT)
3. Age ≥ 18 years
4. ECOG Performance 0-2
5. No serious concomitant disorders (for example marked reduced respiratory capacity, active infection, unstable cardiovascular disease, renal dysfunction) that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study procedure
6. No contraindication for study specific procedure - bronchoscopy, CT, MRI and PET.
7. No conditions - medical, social, psychological - which could prevent adequate information and follow-up
8. No pregnancy or lactating women
9. Written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Progression free survival in one year

CONTACTS AND LOCATIONS:
Overall Officials: Sveinung Sørhaug, MD PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Trondheim University Hospital, Dept of Thoracic Medicine, Trondheim, Norway